CLINICAL TRIAL: NCT06815068
Title: Effect of Simplified Implant Placement Protocols on Failure Rate
Status: Active, not recruiting | Type: Observational
Sponsor: Chrysalis Dental Center (Other)
Responsible Party: Sponsor
Other Study IDs: 00046435
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Dental Implant Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients receiving dental implants: No exclusion criteria

SUMMARY:
The primary objective of this study is to evaluate the effectiveness of implant treatment in an unselected patient population as measured through implant failure.

ELIGIBILITY:
Inclusion Criteria:

* edentulism

Exclusion Criteria:

* ASA class 4

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients requiring dental implants
Sampling Method: Non-Probability Sample
Enrollment: 2700 (Actual)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Implant failure rate | implant placement between 2011 and 2023

CONTACTS AND LOCATIONS:
Locations (1):
- Chrysalis Dental Center, North York, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided